CLINICAL TRIAL: NCT01993459
Title: A Randomized Controlled Trial on the Effects of Midazolam on the Quality of Postoperative Recovery in Patients
Brief Title: The Effects of Midazolam on the Quality of Postoperative Recovery
Acronym: WOLII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Stefan van Beek, BSc, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14091991
Record Dates: First submitted 2013-10-29; First posted 2013-11-25 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Postoperative Period; Anxiety; Fatigue; Depression; Aggression
Keywords: Quality of Recovery
MeSH Terms: conditions — Anxiety Disorders; Fatigue; Depression; Aggression | interventions — Midazolam; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam intravenous (Experimental): 3mg/ml midazolam given intravenously
  Interventions: Drug: Midazolam
- NaCl (sodium chloride) 0,9% (Placebo Comparator): NaCl (sodium chloride) 0,9% given intravenously 3ml.
  Interventions: Drug: NaCl (sodium chloride) 0,9%

INTERVENTIONS:
Drug: Midazolam — We will administer Midazolam 3mg intravenously once pre-operatively to patients just before they undergo surgery
  Other Names: Dormicum
  Arms: Midazolam intravenous
Drug: NaCl (sodium chloride) 0,9% — We will administer NaCl (sodium chloride) 0,9% 3ml intravenously once pre-operatively to patients just before they undergo surgery
  Other Names: saline solution; sodium chloride solution
  Arms: NaCl (sodium chloride) 0,9%

SUMMARY:
The purpose of this study is to determine whether Midazolam given pre-operatively to patients undergoing abdominal surgery improves the quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* All patiënts operated with a laparotomy in the Erasmus Medical Center of Rotterdam, older than 18 years and planned for a postoperative stay for a minimum of 3 days

Exclusion Criteria:

* Pregnant, benzodiazepine usage, contra-indication for midazolam, mental retardation, non-dutch speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Recovery (QoR-40 Scale) | baseline, workday 3 postoperative, workday 7 postoperative

SECONDARY OUTCOMES:
Change in anxiety measured with a Dutch translated State-Trait Anxiety Inventory (STAI) | baseline, workday 1 postoperative, workday 7 postoperative
Change in depressive moods and anxiety measured by a Dutch translation of the Hospital Anxiety and Depression Scale (HADS) | baseline, workday 1 postoperative, workday 7 postoperative
Change in fatigue measured by a validated Dutch questionnaire Multidimensional Fatigue Index : "Multidimensionele Vermoeidheids Index" (MVI-20) | baseline, workday 7 postoperative
Change in self-efficacy measured by a Dutch translation of General Self-Efficacy- Schwarzer (GSES). | baseline, workday 7 postoperative
Change in Systolic bloodpressure | baseline, workday 1 postoperative
Change in self-esteem measured by a Dutch translation of the and Rosenberg self-esteem scale (RSES) | baseline, workday 7 postoperative
Change in Diastolic Blood pressure | baseline, workday 1 postoperative
Temperature after surgery measured with an ear thermometer | directly after surgery
Change in Heart Rate | preoperatively, during surgery and postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jan Stolker, MD, PhD, Study Chair — Erasmus MC Rotterdam Anesthesiology; Markus Klimek, MD, PhD, Study Chair — Erasmus MC Rotterdam Anesthesiology; Stefan van Beek, BSc, Principal Investigator — Erasmus MC Rotterdam Anesthesiology
Locations (1):
- Erasmus Medical Centre, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] van Beek S, Kroon J, Rijs K, Mijderwijk HJ, Klimek M, Stolker RJ. The effect of midazolam as premedication on the quality of postoperative recovery after laparotomy: a randomized clinical trial. Can J Anaesth. 2020 Jan;67(1):32-41. doi: 10.1007/s12630-019-01494-6. Epub 2019 Oct 1. PMID 31576513